CLINICAL TRIAL: NCT05913700
Title: Estimation of Prevalence of and Risk Factor for Respiratory Viruses Among Emergently Admitted Adult Patients With Respiratory Symptoms and Their Influence on Clinical Outcomes in the Settings From Rural to Urban Community Hospitals
Brief Title: Effect of Respiratory Virus Infection on EmeRgencY Admission Study (EVERY Study)
Acronym: EVERY
Status: Active, not recruiting | Type: Observational
Sponsor: Institute for Clinical Effectiveness, Japan (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: ICE_2023_01C
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus (RSV); Respiratory Viral Infection; Acute Disease
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Study design is multicenter prospective registry study. Participants are consecutive (non-selected, a sequential registration) patients admitted from emergency rooms of participating hospitals who meet the eligibility criteria.

The primary objectives are to estimate the prevalence of and risk factors for RS and other respiratory virus infection and their effect on hospital course in patients with any respiratory symptom who admit from emergency room using a multicenter prospective registry study. The primary target virus is RS virus and the secondary target viruses are respiratory virus and other microorganisms measured by FilmArray 2.1.

DETAILED DESCRIPTION:
The investigators register consecutive patients who meet the eligibility criteria at 3 participating hospitals from electronic medical records. As a routine clinical practice, presence of respiratory symptoms using standard electronic medical record (EMR) format are universally assessed at the emergency room when the patients are determined to be admitted. Patients are registered if they meet the eligibility criteria and information of medical history, baseline characteristics, living status, physical findings, laboratory tests, chest X-ray, electrocardiogram, on admission are retrieved from the EMRs. The nasopharyngeal swab is obtained within 24 hours after admission as a standard practice, which will be sampled at either emergency rooms or hospital wards. The swab is transferred to the onsite laboratory office to measure the FilmArray 2.1 by trained technicians or physicians in charge.

Serum antibodies for RS virus are obtained from patients with suspected lower respiratory infection (bronchitis and pneumonia) who provided their written informed consent, at the timing of admission and 4 weeks after the admission.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older
* Admission from emergency room
* Having at least one of following respiratory symptoms/signs for at least 24 hours and the onset date of first symptom/sign less than 7 days before admission, which meet the acute respiratory infection (ARI) case definition described below: nasal congestion, rhinorrhea, sore throat, cough, sputum, dyspnea, wheeze, crackles or rhonchi, tachypnea (>=20 per minute), decreased saturation of oxygen (< 95%), admission with oxygen supplementation

Exclusion Criteria:

* Scheduled admission
* Admission for trauma care
* With nasopharyngeal cavity diseases or deformity which block the nasopharyngeal sampling
* Admission for end of life
* Decline to participate the study by either informed consent or opt-out method

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive (non-selected, a sequential registration) patients admitted from emergency rooms of participating hospitals who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3067 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
RS virus infection | On admission
  Presence of RS virus infection measured by FilmArray 2.1

SECONDARY OUTCOMES:
Respiratory virus and other microorganisms | On admission
  Presence of respiratory virus and other microorganisms measured by FilmArray 2.1
RS virus infection measured by paired serologic tests | 4 weeks
  Presence of RS virus infection measured by paired serologic tests (neutralizing antibody method)
Lower respiratory tract infections | On admission
  Presence of at least 2 lower respiratory symptoms/signs for at least 24 hours including at least 1 lower respiratory sign or presence of at least 3 lower respiratory symptoms for at least 24 hours according to the Table S2 from the following reference.
  Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
All-cause mortality | 30 days
  All-cause mortality
All-cause mortality | 180 days
  All-cause mortality
All-cause readmission | 180 days
  All-cause readmission
Length of hospital stay | 30 days
  Length of hospital stay
Changes in clinical frailty scale | 30 days
  The clinical frailty scale is scored from 1 (very fit) to 9 (terminally ill) according to the following reference.
  Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ 2005;173:489-95
Changes in functional oral intake score | 30 days
  The functional oral intake score is scored from 1 (nothing by mouth) to 7 (total oral diet with no restriction) according to the following reference.
  Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil 2005;86:1516-20
Changes in modified Rankin Scale | 30 days
  The modified Rankin Scale is scored from 0 (no symptoms) to 6 (death) according to the following reference.
  van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke 1988;19:604-7
Presence of nasal congestion or rhinorrhea | 30 days
  Presence of nasal congestion or rhinorrhea is defined by the Table S2 from the following reference.
  Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of sore throat | 30 days
  Presence of sore throat is defined by the Table S2 from the following reference.
  Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of cough | 30 days
  Presence of cough is defined by the Table S2 from the following reference. Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of sputum | 30 days
  Presence of sputum is defined by the Table S2 from the following reference. Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of dyspnea | 30 days
  Presence of dyspnea is defined by the Table S2 from the following reference. Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of wheeze | 30 days
  Presence of wheeze is defined by the Table S2 from the following reference. Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of crackles or rhonchi | 30 days
  Presence of crackles or rhonchi is defined by the Table S2 from the following reference.
  Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Presence of tachypnea | 30 days
  Tachypnea is defined as respiratory rate ≥20 respirations/minute.
Presence of decreased oxygen saturation | 30 days
  Decreased oxygen saturation is defined as <95% or ≤90% if baseline oxygen saturation is <95%.
Presence of oxygen supplementation | 30 days
  Oxygen supplementation is any supplementation of oxygen including nasal, nasal high-flow supply, oxygen mask, ventilator, or extracorporeal membrane oxygenation.
Length from onset to admission of acute respiratory infection symptoms | 7 days
  Length from onset to admission of acute respiratory infection symptoms
Presence of family member who attends preschool or school | On admission
  Presence of family member who attends preschool or school
Presence of symptoms of family member | On admission
  Family member is defined as those who live with the patient. Symptoms include fever, nasal congestion, rhinorrhea, sore throat, cough, sputum, dyspnea, or wheeze according to the Table S2 from the following reference.
  Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrøm V; AReSVi-006 Study Group. Respiratory syncytial virus prefusion F protein vaccine in older adults. N Engl J Med 2023;388:595-608
Use of antimicrobials | 30 days
  Use of any antimicrobials during the hospital stay
Admission to intensive or high care unit | 30 days
  Admission to intensive or similar high care unit
Respiratory complications | 30 days
  Each of following respiratory complications is separately assessed: pneumonia, respiratory failure, fever
Cardiovascular complications | 30 days
  Each of following cardiovascular complications is separately assessed: ischemic heart diseases, atrial fibrillations, valvular heart disease, heart failure necessitating drug therapy, deep venous thromboembolism or pulmonary embolism, peripheral artery disease necessitating drug therapy, hypertension necessitating drug therapy
Cerebrovascular complications | 30 days
  Each of following cerebrovascular complications is separately assessed: ischemic stroke (excluding transient ischemic attack), intracranial hemorrhage, subarachnoid hemorrhage

OTHER OUTCOMES:
Number of safety outcome | 4 weeks
  Insert site bleeding or peripheral nerve injury by blood drawing
Number of any adverse events | 180 days
  Any adverse events which are considered to be related to the study by site investigators

CONTACTS AND LOCATIONS:
Overall Officials: Tsukasa Nakamura, MD, PhD, Principal Investigator — Shimane Prefectural Central Hospital
Locations (3):
- Japan (3):
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Nara City Hospital, Nara, Nara
  - Shimane Prefectural Central Hospital, Izumo, Shimane

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morimoto T, Morikawa T, Imura H, Nezu M, Hamazaki K, Sakuma M, Chaumont A, Moitinho de Almeida M, Moreno VP, Ho Y, Harrington L, Matsuki T, Nakamura T. Rationale and protocol for a prospective cohort study of respiratory viral infections in patients admitted from emergency departments of community hospitals: Effect of respiratory Virus infection on EmeRgencY admission (EVERY) study. BMJ Open. 2024 Apr 15;14(4):e081037. doi: 10.1136/bmjopen-2023-081037. PMID 38626982